CLINICAL TRIAL: NCT03214978
Title: Targeted-sequencing of PTC in Different Stages
Acronym: PTC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, LI Yi, Doctor, Shanghai 6th People's Hospital
Other Study IDs: LY-US-THY-001
Record Dates: First submitted 2017-07-11; First posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Exploratory Study
Keywords: thyroid
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prevalence of papillary thyroid micro-carcinoma (PTMC) increased rapidly in recent years but the design of treatment is controversial because a majority of them are indolent. Therefore, to recognize which PTMC is of strong progressive potential which should be operated is very crucial. Fine needle aspiration (FNA) pre-surgery could obtain tumor cells which could be used in genetic analysis. To date, there is no specific way to evaluate the aggressive potential of a PTMC pre-surgery. So, the purpose of this proposal is to screen genetic mutations of the aggressive type of PTMC. The candidate did a whole exome sequencing on 3-3 pairs of PTCs and found some SNPs and Indels in TP53、TTN、PDF. To further investigate those mutations, a target region sequencing will be done in 40 pairs tumor samples. And ultimately to find out which genetic event could contribute to strong aggressive potential of PTC. The mutations details would be design to test the FNA and tissue sample to validate if the genetic testing based on FNA is reliable. The gene test results would be evaluated with sonographic features to predict the potential of small thyroid carcinoma before surgery. This project won't aim to study the function and mechanism of specific genes but just screen them out. So, the fund would cover the fee of the whole study and this study is very likely to achieve the goal.

ELIGIBILITY:
Inclusion Criteria:

* patients who will receive thyroid resection

Exclusion Criteria:

* patients who has been radiologically treated

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: DNA will be extracted from of 40 pairs tumor samples including 40 patients in 4 groups (stage I, II, III and IV)
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-07-30 (Estimated); Primary Completion 2017-12-01 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
types of mutation of targets genes in papillary thyroid carcinomas in different stages | 2018-1-1
  types of mutation of targets genes in papillary thyroid carcinomas in different stages